CLINICAL TRIAL: NCT00903370
Title: Surgical Ablation Versus No Surgical Ablation for Patients With Persistent or Longstanding Persistent Atrial Fibrillation (AF) Undergoing Mitral Valve Surgery
Brief Title: Surgical Ablation Versus No Surgical Ablation for Patients With Atrial Fibrillation Undergoing Mitral Valve Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annetine Gelijns (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Annetine Gelijns, Professor of Health Policy, Chair Department of Health Evidence & Policy, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 08-1078-0004; U01HL088942 (NIH); U01HL088942-03 (NIH); 656 (Other: Cardiothoracic Surgical Trials Network)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation; Mitral Valve Insufficiency; Mitral Valve Stenosis
Keywords: Mitral Valve Regurgitation; Mitral Valve Surgery; Mitral Valve Disease; Ablation, Catheter; Catheter Ablation, Radiofrequency
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Insufficiency; Mitral Valve Stenosis | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MVS (Active Comparator): All participants will undergo mitral valve surgery with ligation/excision of left atrial appendage.
  Interventions: Procedure: MVS
- Ablation (Experimental): Participants will undergo mitral valve surgery with ligation/excision of left atrial appendage plus surgical ablation with pulmonary vein isolation or biatrial lesion set.
  Interventions: Procedure: MVS; Device: Ablation

INTERVENTIONS:
Procedure: MVS — All participants will have their left atrial appendage excised or excluded. For mitral regurgitation, the procedures will be a valve repair in the majority of cases. For valves that are not amenable to repair, and for most cases of mitral stenosis, a valve replacement will be performed.
  Other Names: Mitral Valve Repair; Mitral Valve Replacement
Device: Ablation — For participants treated by pulmonary vein isolation, two separate encircling lesions will be made around the left and right pulmonary veins. For participants treated with biatrial maze lesion set, the left atrial lesions will include, the two encircling lesions, as well as connecting lesions between to the pulmonary veins, from the pulmonary veins to the mitral valve annulus, and from the pulmonary veins to the left atrial appendage. The right pulmonary veins will be isolated first. Isolation will be confirmed by pacing the pulmonary veins at the previously identified threshold for capture. If no atrial capture is noted, it will be inferred that the right pulmonary veins were isolated. If atrial capture is noted, additional ablations on the atrial cuff will be performed until isolation is confirmed. This will be repeated on the left pulmonary veins.
  Other Names: Surgical Ablation
  Arms: Ablation

SUMMARY:
The purpose of the research is to determine whether treating atrial fibrillation with surgical ablation during scheduled mitral valve surgery is better than mitral valve surgery by itself without the surgical ablation. Surgical ablation of atrial fibrillation is a technique used by surgeons to deaden atrial heart tissue and block electrical signals that may be causing your heart to beat irregularly. There are no new procedures being tested in this study; both mitral valve surgery and surgical ablation are used regularly in patients who have mitral valve problems and atrial fibrillation, although no surgical ablation devices have been approved by the Food and Drug Administration for the treatment of atrial fibrillation. What is not known with certainty, is whether patients with atrial fibrillation who are having planned mitral valve surgery would do better if they also had surgical ablation rather than medication alone to treat their atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the addition of surgical ablation to planned mitral valve surgery for patients with persistent or longstanding persistent AF (within 6 months prior to randomization) reduces the incidence of postoperative heart arrhythmia compared to mitral valve repair with medication therapy alone. This is a randomized, multi-center trial which will enroll 260 subjects who will be randomized in a 1:1 fashion to: (a) mitral valve surgery plus surgical ablation or (b) mitral valve surgery without ablation (control group). All patients will undergo ligation or excision of the left atrial appendage. Patients assigned to the ablation group will be further randomized (1:1) to one of two lesion sets: (1) pulmonary vein isolation only or (2) biatrial Maze lesions. The target population for this trial consists of adult patients with mitral valve disease requiring surgical intervention and persistent or longstanding persistent atrial fibrillation. All patients who meet the eligibility criteria may be included in the study regardless of gender, race or ethnicity. The primary efficacy endpoint is freedom from AF, which will be measured by 3-day continuous monitoring at 6 months and 12 months post-ablation. The primary safety endpoint is a composite of death, stroke, serious cardiac events (heart failure, myocardial infarction), cardiac re-hospitalizations, transient ischemic attack, pulmonary embolism, peripheral embolism, excessive bleeding, deep sternal wound infection/mediastinitis, damage to specialized conduction system requiring permanent pacemaker, damage to peripheral structures, such as the esophagus, within 30 days post-procedure or hospital discharge (whichever is later).

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age ≥ 18 years
* Clinical indications for mitral valve surgery for the following:

  1. Organic mitral valve disease; or
  2. Functional non-ischemic mitral regurgitation; or
  3. Ischemic mitral regurgitation with evidence of concomitant structural mitral valve disease

Note: May include need for surgical management of functional tricuspid regurgitation or patent foramen ovale. May also include concomitant CABG, aortic arch or aortic valve procedure. Surgical intervention may be performed via sternotomy or minimally invasive procedure.

* a) Persistent AF within 6 months prior to randomization, defined as non self-terminating AF lasting greater than 7 days but no more than one year, or lasting less than 7 days but necessitating pharmacologic or electrical cardioversion.

  * Duration of AF must be documented by medical history and
  * Presence of AF must be documented by a direct electrocardiographic assessment within 6 months prior to randomization.
* b) Longstanding persistent AF is defined as continuous AF of greater than one year duration.

  * Duration of AF must be documented by medical history and
  * Presence of AF must be documented by a direct electrocardiographic assessment upon arrival in the OR.
* Able to use heart rhythm monitor

Exclusion Criteria:

* 1. AF without indication for mitral valve surgery 2. AF is paroxysmal 3. Evidence of left atrial thrombus by intra-operative TEE 4. Evidence of active infection 5. Mental impairment or other conditions that may not allow subject to understand the nature, significance, and scope of study 6. Surgical management of hypertrophic obstructive cardiomyopathy 7. Previous catheter ablation for AF 8. Life expectancy of less than one year 9. Absolute contraindications for anticoagulation therapy 10. Enrollment in concomitant drug or device trials 11. Uncontrolled hypo- or hyperthyroidism 12. FEV1 < 30% of predicted value and/or need for home oxygen therapy 13. Women who are pregnant as evidenced by positive pregnancy test 14. Women of childbearing age who do not agree to be on adequate birth control throughout the period of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gardner, MD, Study Chair — Christiana Care Health Services; Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital; Annetine C. Gelijns, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (21):
- United States (18):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Montreal Heart Institute, Montreal, Quebec
  - Quebec Heart Institute/Laval Hopital, Québec, Quebec

REFERENCES:
- [Result] Gillinov AM, Gelijns AC, Parides MK, DeRose JJ Jr, Moskowitz AJ, Voisine P, Ailawadi G, Bouchard D, Smith PK, Mack MJ, Acker MA, Mullen JC, Rose EA, Chang HL, Puskas JD, Couderc JP, Gardner TJ, Varghese R, Horvath KA, Bolling SF, Michler RE, Geller NL, Ascheim DD, Miller MA, Bagiella E, Moquete EG, Williams P, Taddei-Peters WC, O'Gara PT, Blackstone EH, Argenziano M; CTSN Investigators. Surgical ablation of atrial fibrillation during mitral-valve surgery. N Engl J Med. 2015 Apr 9;372(15):1399-409. doi: 10.1056/NEJMoa1500528. Epub 2015 Mar 16. PMID 25853744
- [Derived] DeRose JJ Jr, Mancini DM, Chang HL, Argenziano M, Dagenais F, Ailawadi G, Perrault LP, Parides MK, Taddei-Peters WC, Mack MJ, Glower DD, Yerokun BA, Atluri P, Mullen JC, Puskas JD, O'Sullivan K, Sledz NM, Tremblay H, Moquete E, Ferket BS, Moskowitz AJ, Iribarne A, Gelijns AC, O'Gara PT, Blackstone EH, Gillinov AM; CTSN Investigators. Pacemaker Implantation After Mitral Valve Surgery With Atrial Fibrillation Ablation. J Am Coll Cardiol. 2019 May 21;73(19):2427-2435. doi: 10.1016/j.jacc.2019.02.062. PMID 31097163
- See also: Click here for the Cardiothoracic Surgical Trials Network Web site — http://www.ctsurgerynet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- MVS Alone: Participants will undergo mitral valve surgery with ligation/excision of left atrial appendage.
  MVS alone: All participants will have their left atrial appendage excised or excluded. For mitral regurgitation, the procedures will be a valve repair in the majority of cases. For valves that are not amenable to repair, and for most cases of mitral stenosis, a valve replacement will be performed.
- MVS + Ablation: Participants will undergo mitral valve surgery with ligation/excision of left atrial appendage plus surgical ablation with pulmonary vein isolation or biatrial lesion set.
  MVS + ablation: For participants treated by pulmonary vein isolation, two separate encircling lesions will be made around the left and right pulmonary veins.
  For participants treated with biatrial maze lesion set, the left atrial lesions will include the two encircling lesions, as well as connecting lesions between to the pulmonary veins, from the pulmonary veins to the mitral valve annulus, and from the pulmonary veins to the left atrial appendage. The right pulmonary veins will be isolated first. Isolation will be confirmed by pacing the pulmonary veins at the previously identified threshold for capture. If no atrial capture noted, it will be inferred that the right pulmonary veins were isolated. If atrial capture noted, additional ablations on the atrial cuff will be performed until isolation is confirmed.
Period: Overall Study
Arm/Group | MVS Alone | MVS + Ablation
Started | 127 | 133
Completed | 99 | 109
Not Completed | 28 | 24
Not completed — Death | 13 | 10
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVS Alone | MVS + Ablation | Total
Number analyzed (Participants) | 127 | 133 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (10) | 69.7 (10.4) | 69.6 (10.2)
Gender [Count of Participants; unit: Participants]
  Female | 63 | 57 | 120
  Male | 64 | 76 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 119 | 123 | 242
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 112 | 116 | 228
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 22 | 43
  United States | 106 | 111 | 217

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Atrial Fibrillation
Time Frame: Measured at Month 12
Population: Since the primary analysis is an intent-to-treat, outcomes were imputed for patients with missing data.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | MVS Alone | MVS + Ablation
Number analyzed (Participants) | 127 | 133
percentage of patients | 31.1 [22.6 to 40.1] | 61.8 [51.4 to 72.2]

2. Secondary Outcome: Composite of Death, Stroke, Serious Adverse Events (Cardiac and Non-cardiac), and Cardiac Re-hospitalizations Less Than 30 Days Post-procedure or Hospital Discharge
Time Frame: Less than 30 days post-procedure or hospital discharge
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | MVS Alone | MVS + Ablation
Number analyzed (Participants) | 127 | 133
percentage of patients | 22.8 [15.5 to 30.1] | 31.6 [23.7 to 39.5]

ADVERSE EVENTS:
Arm/Group | MVS Alone | MVS + Ablation
Serious Adverse Events (participants affected / at risk) | 69/127 | 77/133
Other Adverse Events (participants affected / at risk) | 36/127 | 40/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVS Alone (N=127) | MVS + Ablation (N=133)
Bleeding (General disorders) | 6 (6) | 7 (7)
Arrhythmias-Sustained ventricular arrhythmia (Cardiac disorders) | 6 (6) | 4 (4)
Arrhythmias-Sustained supraventricular arrhythmia (Cardiac disorders) | 16 (21) | 19 (30)
Cardiac conduction abnormalities requiring PPM (Cardiac disorders) | 9 (9) | 25 (25)
Pericardial Fluid Collection (Cardiac disorders) | 5 (5) | 4 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Non-infectious Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hepatic Dysfunction (Hepatobiliary disorders) | 3 (3) | 3 (3)
Major Infection - Localized - Pneumonia (Infections and infestations) | 10 (11) | 3 (3)
Major Infection - Localized - Other (Infections and infestations) | 7 (7) | 8 (10)
Major Infection - Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Major Infection - Sepsis (Infections and infestations) | 4 (4) | 8 (8)
Heart Failure (Cardiac disorders) | 11 (13) | 14 (19)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 2 (2)
Neurological Dysfunction - CVA-Ischemic (Nervous system disorders) | 3 (3) | 3 (4)
Neurological Dysfunction - CVA-Hemorrhagic (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neurological Dysfunction - Other (not stroke, TIA, Toxic Metabolic Encephalopathy) (Nervous system disorders) | 1 (1) | 3 (3)
Renal Dysfunction (no dialysis) (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal Failure (dialysis) (Renal and urinary disorders) | 2 (2) | 4 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 6 (6)
Right Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Venous Thromboembolism Event (Vascular disorders) | 3 (4) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVS Alone (N=127) | MVS + Ablation (N=133)
Bleeding (General disorders) | 0 (0) | 2 (2)
Arrhythmias-Sustained supraventricular arrhythmia (Cardiac disorders) | 15 (19) | 11 (12)
Cardiac conduction abnormalities requiring PPM (Cardiac disorders) | 3 (3) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Major Infection - Localized - Other (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Neurological Dysfunction - Toxic Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Neurological Dysfunction - Other (not stroke, TIA, Toxic Metabolic Encephalopathy) (Nervous system disorders) | 2 (2) | 2 (2)
Renal Dysfunction (no dialysis) (Renal and urinary disorders) | 2 (2) | 3 (3)
Venous Thromboembolism Event (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No